CLINICAL TRIAL: NCT01044147
Title: Online Counseling to Enable Lifestyle-focused Obesity Treatment in Primary Care
Acronym: OCELOT-PC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathleen McTigue, Assitant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R18HS018155 (AHRQ)
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: Obesity; Internet
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VLM-S (Experimental): Participants in this arm receive "standard" lifestyle coaching, which is delivered on a specified schedule. They will also receive online information about evidence-based lifestyle goals and links to reputable resources for helping to achieve a healthy lifestyle.
  Interventions: Behavioral: VLM-S
- VLM-M (Experimental): Participants in this arm receive "modulated" lifestyle coaching, where coaching frequency may be adjusted according to whether the participant is meeting program goals for program use and targeted behaviors. They will also receive online information about evidence-based lifestyle goals and links to reputable resources for helping to achieve a healthy lifestyle.
  Interventions: Behavioral: VLM-M
- OGR (Active Comparator): Participants in this arm will receive online information about evidence-based lifestyle goals and links to reputable resources for helping to achieve a healthy lifestyle, but not personalized lifestyle coaching.
  Interventions: Behavioral: OGR

INTERVENTIONS:
Behavioral: VLM-S — Online program for weight loss - standard
  Arms: VLM-S
Behavioral: VLM-M — Online program for weight loss - modulated
  Arms: VLM-M
Behavioral: OGR — Online program for weight loss - resources
  Arms: OGR

SUMMARY:
With over half of the US population currently overweight and 31% of adults now obese, the primary care setting may represent an important source of weight-loss support, in the interest of cardiovascular prevention. Yet, although the US Preventive Services task force recommends that physicians screen all adult patients for obesity and offer intensive counseling and behavioral interventions to promote sustained weight loss for obese adults, the recommendation has not been widely implemented. The Internet may help overcome many of the barriers that have prevented intensive obesity counseling in the clinical setting. The aim of this study is to examine whether Internet-based interventions for developing healthier lifestyles can improve preventive health care in a cost-effective manner.

DETAILED DESCRIPTION:
The study, Online counseling to enable lifestyle-focused obesity treatment in primary care, aims to translate an evidence-based lifestyle intervention into the primary care setting, using information technology to enable clinical lifestyle counseling. While the US Preventive Services Task Force (USPSTF) recommends that clinicians screen all adult patients for obesity and offer intensive counseling and behavioral interventions to promote sustained weight loss for obese adults, multiple barriers to intensive lifestyle counseling exist and the recommendation has not been widely implemented. By requiring physician referral, augmenting the health care team's access to behavioral expertise, and encouraging physician feedback to participating patients, we aim to integrate lifestyle issues into routine preventive medicine. We will examine change in weight, waist circumference, physical activity, quality of life, and will calculate intervention cost-effectiveness. We will ensure sustainability by using recruitment and adherence strategies that can be replicated in routine practice, and counseling staff who are representative of the educators employed in primary care practice. If an online strategy is effective, the extensive network of the University of Pittsburgh Medical Center Health System provides excellent infrastructure for supporting dissemination in the region. As such, this study may facilitate wide-spread adoption of current evidence-based preventive medicine guidelines recommending incorporation of intensive lifestyle interventions into primary care practice.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI > 30kg/meters squared)
* Age 21-75
* Receives primary care at a participating primary care clinic in the Pittsburgh, PA area

Exclusion Criteria:

* Primary care physician determination that moderate physical activity is not safe or appropriate for the patient
* Pregnancy
* Planned pregnancy in the next 2 years
* Current breast-feeding
* Bariatric surgery in the past 2 years
* Planned bariatric surgery in the next 2 years
* Edematous state that interferes with body weight assessment
* Health condition that is likely to influence body weight
* Heart attack within the past 3 months
* Regular use of prescription medication that is likely to influence body weight
* participation during the past year in either of the pilot programs for this study
* perceived lack of basic computer or Internet skills
* Inability to learn adequately from English language audio-recorded materials
* Lack of access to a scale
* Inability to attend an Orientation session

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in body weight (Kg) | 1 year

SECONDARY OUTCOMES:
% obtaining >7% weight loss | 1 year
Change in BMI (kg/m2) | 1 year
Change in waist circumference | 1 year
Change in steps per day | 1 year
Change in health-related quality of life as measured by the RAND-36 PCS or MCS | 1 year
Change in total score on IWQol-Lite | 1 year
% with >70 meter increase on 6-minute walk | 1 year
Change in blood pressure (mm Hg) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M McTigue, MD, MS, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Diabetes Prevention Program (DPP) Research Group. The Diabetes Prevention Program (DPP): description of lifestyle intervention. Diabetes Care. 2002 Dec;25(12):2165-71. doi: 10.2337/diacare.25.12.2165. PMID 12453955